CLINICAL TRIAL: NCT02251327
Title: Feasibility and Accuracy of a Novel Xpert Cartridge for Rapid Molecular Detection of Drug Resistant Mycobacterium Tuberculosis in Sputum
Brief Title: Feasibility and Accuracy of a Novel Xpert Cartridge
Acronym: (XpertDST)
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NA_0008420; NA_0008420 (Other: Johns Hopkins University)
Record Dates: First submitted 2014-09-23; First posted 2014-09-29 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case detection group: Suspected or confirmed new pulmonary tuberculosis cases who have received anti-tuberculosis drugs for less than 3 (three) days and provide up to two expectorated sputum specimens. One investigational Xpert DST test and one Xpert MTB/RIF test were performed directly on the same sputum specimen; in addition, one smear microscopy test, one mycobacterial liquid culture, and one solid culture were performed after digestion and decontamination of sputum.
  Interventions: Device: Investigational Xpert DST test
- Drug resistance risk group: Confirmed pulmonary tuberculosis cases with documented rifampin resistance, who have received anti-tuberculosis drugs for 31 days or less and/or history of prior tuberculosis PLUS ongoing signs and/or cases with symptoms of pulmonary tuberculosis PLUS suspected drug resistance and provide up to two expectorated sputum specimens. One investigational Xpert DST test and one Xpert MTB/RIF test were performed directly on the same sputum specimen; in addition, one smear microscopy test, one mycobacterial liquid culture, and one solid culture were performed after digestion and decontamination of sputum.
  Interventions: Device: Investigational Xpert DST test

INTERVENTIONS:
Device: Investigational Xpert DST test — One investigational test performed directly on the same sputum specimen.

SUMMARY:
Consenting adults will be interviewed for demographic and medical information, and then will be asked to provide two expectorated sputum specimens. In the study laboratory, sputa will be tested using conventional and investigational diagnostic tests for tuberculosis.

DETAILED DESCRIPTION:
* For each of isoniazid, ofloxacin, moxifloxacin, amikacin, and kanamycin: sensitivity and specificity of the investigational Xpert test for detection of drug resistance, using phenotypic drug susceptibility testing as the reference comparator
* For each of isoniazid, ofloxacin, moxifloxacin, amikacin, and kanamycin: sensitivity and specificity of the investigational Xpert test for detection of drug resistance, using mycobacterial DNA sequencing as the reference comparator
* Sensitivity and specificity, for detection of M. tuberculosis in sputum, of the investigational Xpert test and of the conventional Xpert MTB/RIF test, using culture as the reference comparator
* Diagnostic yield (for tuberculosis) of the investigational Xpert test and of the conventional Xpert MTB/RIF test
* For the investigational Xpert test, the proportion of specimens with a result of 'invalid' and the proportion of specimens with a result of 'error'
* Proportion of study participants with M. tuberculosis detected in sputum
* Proportion of participants with drug resistant tuberculosis, by drug resistance pattern and by tuberculosis categorization (new case or not new case)

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all of the following inclusion criteria in order to be eligible to participate:

  * Age ≥ 19 years (age of majority) if enrolled in South Korea; age ≥ 18 years (age of majority) if enrolled in China
  * Provision of informed consent
  * Clinical signs and/or symptoms suggestive of pulmonary tuberculosis
  * Meets one of the following criteria:

A. Suspected or confirmed new pulmonary tuberculosis case who has received anti-tuberculosis drugs for less than 3 (three) days (target enrollment for Group A is approximately 50 participants).

B. Confirmed pulmonary tuberculosis with documented rifampin resistance, who has received anti-tuberculosis drugs for 31 days or less C. History of prior tuberculosis PLUS ongoing signs and/or symptoms of pulmonary tuberculosis PLUS suspected drug resistance

Exclusion Criteria:

* Inability to provide a sputum specimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with clinical signs and/or symptoms of pulmonary TB
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2014-06-04 (Actual); Primary Completion 2015-06-15 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity | 10 months
  sensitivity and specificity of the investigational Xpert DST test for detection of drug resistance, using phenotypic drug susceptibility testing, mycobacterial DNA sequencing, and MTB/RIF test as the reference comparator

SECONDARY OUTCOMES:
Diagnostic yield (for tuberculosis) of the investigational Xpert test and of the conventional Xpert MTB/RIF test | 10 months
the proportion of specimens with a result of 'invalid' and the proportion of specimens with a result of 'error' | 10 months
Proportion of study participants with TB and DRTB | 10 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xie YL, Chakravorty S, Armstrong DT, Hall SL, Via LE, Song T, Yuan X, Mo X, Zhu H, Xu P, Gao Q, Lee M, Lee J, Smith LE, Chen RY, Joh JS, Cho Y, Liu X, Ruan X, Liang L, Dharan N, Cho SN, Barry CE 3rd, Ellner JJ, Dorman SE, Alland D. Evaluation of a Rapid Molecular Drug-Susceptibility Test for Tuberculosis. N Engl J Med. 2017 Sep 14;377(11):1043-1054. doi: 10.1056/NEJMoa1614915. PMID 28902596